CLINICAL TRIAL: NCT01070264
Title: A Pilot Observational Clinical Survey: Impacts of Tahitian Noni Juice on the Quality of Life of Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Excellence in Academic Medicine (EAM) Grant (Unknown)
Responsible Party: Mian-Ying Wang, University of Illinois-Chicago College of Medicine at Rockford
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 20050074
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2007-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noni Juice (Experimental): This was an open label three-month intervention pilot study. Data were collected by pre and post intervention survey as well as laboratory testing. Inclusion criteria were: adults of both sexes aged 40 to 75, with a diagnosis of OA on the hip or knee by their primary care physician, not on prescription medicine for OA, and who were willing to drink 3 oz of TNJ a day
  Interventions: Dietary Supplement: Noni Juice

INTERVENTIONS:
Dietary Supplement: Noni Juice — This was an open label three-month intervention pilot study. Data were collected by pre and post intervention survey as well as laboratory testing. Inclusion criteria were: adults of both sexes aged 40 to 75, with a diagnosis of OA on the hip or knee by their primary care physician, not on prescription medicine for OA, and who were willing to drink 3 oz of TNJ a day

SUMMARY:
Tahitian Noni Juice (TNJ) made from Morinda citrifolia (noni) fruits may provide a safe adjunctive treatment for osteoarthritis (OA) due to its anti-inflammatory and analgesic properties. In this study the investigators examined whether TNJ was able to improve the symptoms and quality of life (QOL) of OA patients. The investigators also sought to evaluate the tolerability and safety of TNJ.

This was an open label three-month intervention pilot study. Data were collected by pre and post intervention survey as well as laboratory testing. Inclusion criteria were: adults of both sexes aged 40 to 75, with a diagnosis of OA on the hip or knee by their primary care physician, not on prescription medicine for OA, and who were willing to drink 3 oz of TNJ a day.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 40 to 75 of both sexes with a physician diagnosis of OA of the hip or knee who were not taking prescription medicine for arthritis and were willing to drink 3 oz of TNJ daily for 12 weeks

Exclusion Criteria:

* all others

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois-Chicago College of Medicine at Rockford, Rockford, Illinois, United States